CLINICAL TRIAL: NCT03968809
Title: Role of the Cardioflux Magnetocardiography System in Predicting Patient Outcomes With Coronary Artery Disease
Brief Title: Role of Cardioflux in Predicting Coronary Artery Disease (CAD) Outcomes
Status: Completed | Type: Observational
Sponsor: Genetesis Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: 1902469303
Record Dates: First submitted 2019-05-28; First posted 2019-05-30 (Actual); Last update posted 2023-02-23 (Actual); Status verified 2023-02

CONDITIONS: Coronary Artery Disease
Keywords: Coronary Artery Disease; Cardiac Imaging
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Standard Coronary Artery Disease Screening: All patients presenting for standard coronary artery disease screening will undergo additional imaging with CardioFlux MCG. These patients will be followed longitudinally for short and long term MACE.
  Interventions: Diagnostic Test: CardioFlux Magnetocardiography

INTERVENTIONS:
Diagnostic Test: CardioFlux Magnetocardiography — All patients enrolled and receiving standard screening tests for CAD will undergo a 2 minute scan with MCG. It will be determined if MCG scanning can provide equal or superior accuracy to predict MACE than standard testing.

SUMMARY:
This single-center clinical trial is designed to evaluate the CardioFlux magnetocardiograph diagnostic imaging system to predict major adverse cardiac events (MACE) in patients referred for evaluation for coronary artery disease.

DETAILED DESCRIPTION:
This is a single-center, prospective, observational cohort trial to form a registry data set. Patients presenting for cardiac stress testing utilizing Single Photon Emission Computed Tomography (SPECT), cardiac CT angiography (CCTA), or cardiac catheterization will be offered to enroll in the registry and provide informed consent to undergo imaging with a CardioFlux magnetocardiography (MCG) prior to their procedure.

Multiple studies have shown that MCG accuracy is quite high in identifying patients with symptomatic coronary artery disease. This difference is dramatic enough to prove superiority over standard ECGs in diagnosis of vital ischemic and infarction parameters. Genetesis presents a novel MCG analysis system called CardioFlux (CF). This modality takes less than five minutes to complete, is radiation-free, and is an easy to operate system. This clinical trial will enroll patients of all cardiac risk levels presenting for various modalities of cardiac diagnostic testing to have CardioFlux scanning in addition to standard of care. Results will be interpreted and compared to the immediate results of nuclear (SPECT) stress testing, cardiac CT angiography, or cardiac catheterization.

Participants will be followed up at 30 days and 1 year via phone call or chart review. 30 day and 1 year MACE will be recorded and correlated with initial CardioFlux MCG results. Sensitivity, specificity, positive predictive value (PPV), negative predictive value (NPV), and overall accuracy will be calculated of CardioFlux relative to the incidence of MACE, and in comparison to the above diagnostic modalities.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 years of age at the time of enrollment.
* Patient presenting for cardiac stress testing, cardiac CT angiography (CCTA), or cardiac catheterization.
* Consents to having an magnetocardiogram-CardioFlux study scan.

Exclusion Criteria:

* < 18 years of age
* Patients unable to fit into device
* Non-ambulatory patients
* Patients with implanted cardiac pacemakers/defibrillators
* Positive response on provided Metallic/Ferromagnetic Device Screening Form
* Atrial fibrillation with rapid ventricular response
* Patients with other sustained or incessant arrhythmias
* Patients with claustrophobia or unable to lie supine for 2 minutes
* Patients require supplemental oxygen at home
* Presence or reasonable clinical suspicion of any acute coronary syndrome for which delayed intervention could increase the risk or magnitude of damaged myocardium
* Patients scheduled for cardiac catheterization with indication of valvular disease
* Poor candidate for follow-up (e.g. no access to phone)
* Prisoners
* Repeat participants
* Patients participate in other research studies

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This is an adult patient population at varying risk for coronary artery disease who will present at single center for cardiovascular screening with stress testing, CCTA, or cardiac catheterization with angiography.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2019-09-05 (Actual); Primary Completion 2020-06-20 (Actual); Study Completion 2020-06-20 (Actual)

PRIMARY OUTCOMES:
Percentage study subjects having coronary Revascularization | 1 year
  Patient follow up will be performed to find the incidence of coronary revascularization at 30 days and 1 year.
Percentage of study subjects having Major Adverse Cardiac Events | 1 year
  Patients will have follow up to determine the occurrence of MACE, defined as nonfatal stroke, nonfatal myocardial infarction, and cardiovascular death
Incidence of study subjects with endpoint of death | 1 year
  All cause mortality will be recorded at end of follow up period for the entire study population.

SECONDARY OUTCOMES:
Comparison of MCG with Stress testing | 30 days
  Comparison with nuclear stress testing (SPECT) will be performed, with statistical analysis including sensitivity, specificity, NPV, and PPV
Comparison of MCG with Cardiac CT angiography (CCTA) | 30 days
  Comparison with CCTA will be performed for those having this test, with statistical analysis including sensitivity, specificity, NPV, and PPV

CONTACTS AND LOCATIONS:
Overall Officials: Partho P Sengupta, M.D., Principal Investigator — WVU Heart and Vascular Institute, J.W. Ruby Memorial Hospital
Locations (1):
- J.W. Ruby Memorial Hospital, Morgantown, West Virginia, United States

IPD SHARING:
Plan to Share IPD: No
Currently there is no plan to share independent participant data to other researchers outside the primary institution where the trial is taking place.

REFERENCES:
- [Background] Benjamin EJ, Blaha MJ, Chiuve SE, Cushman M, Das SR, Deo R, de Ferranti SD, Floyd J, Fornage M, Gillespie C, Isasi CR, Jimenez MC, Jordan LC, Judd SE, Lackland D, Lichtman JH, Lisabeth L, Liu S, Longenecker CT, Mackey RH, Matsushita K, Mozaffarian D, Mussolino ME, Nasir K, Neumar RW, Palaniappan L, Pandey DK, Thiagarajan RR, Reeves MJ, Ritchey M, Rodriguez CJ, Roth GA, Rosamond WD, Sasson C, Towfighi A, Tsao CW, Turner MB, Virani SS, Voeks JH, Willey JZ, Wilkins JT, Wu JH, Alger HM, Wong SS, Muntner P; American Heart Association Statistics Committee and Stroke Statistics Subcommittee. Heart Disease and Stroke Statistics-2017 Update: A Report From the American Heart Association. Circulation. 2017 Mar 7;135(10):e146-e603. doi: 10.1161/CIR.0000000000000485. Epub 2017 Jan 25. No abstract available. Erratum In: Circulation. 2017 Mar 7;135(10):e646. doi: 10.1161/CIR.0000000000000491. Circulation. 2017 Sep 5;136(10):e196. doi: 10.1161/CIR.0000000000000530. PMID 28122885
- [Background] Chaikovsky I, Hailer B, Sosnytskyy V, Lutay M, Mjasnikov G, Kazmirchuk A, Bydnyk M, Lomakovskyy A, Sosnytskaja T. Predictive value of the complex magnetocardiographic index in patients with intermediate pretest probability of chronic coronary artery disease: results of a two-center study. Coron Artery Dis. 2014 Sep;25(6):474-84. doi: 10.1097/MCA.0000000000000107. PMID 24667125
- [Background] Goernig M, Liehr M, Tute C, Schlosser M, Haueisen J, Figulla HR, Leder U. Magnetocardiography based spatiotemporal correlation analysis is superior to conventional ECG analysis for identifying myocardial injury. Ann Biomed Eng. 2009 Jan;37(1):107-11. doi: 10.1007/s10439-008-9598-5. Epub 2008 Nov 18. PMID 19015988
- [Background] Kwong JS, Leithauser B, Park JW, Yu CM. Diagnostic value of magnetocardiography in coronary artery disease and cardiac arrhythmias: a review of clinical data. Int J Cardiol. 2013 Sep 1;167(5):1835-42. doi: 10.1016/j.ijcard.2012.12.056. Epub 2013 Jan 19. PMID 23336954
- [Background] Li Y, Che Z, Quan W, Yuan R, Shen Y, Liu Z, Wang W, Jin H, Lu G. Diagnostic outcomes of magnetocardiography in patients with coronary artery disease. Int J Clin Exp Med. 2015 Feb 15;8(2):2441-6. eCollection 2015. PMID 25932186
- [Background] Lim HK, Kwon H, Chung N, Ko YG, Kim JM, Kim IS, Park YK. Usefulness of magnetocardiogram to detect unstable angina pectoris and non-ST elevation myocardial infarction. Am J Cardiol. 2009 Feb 15;103(4):448-54. doi: 10.1016/j.amjcard.2008.10.013. Epub 2008 Dec 25. PMID 19195500
- [Background] Her AY, Park JW. Repolarization Heterogeneity of Magnetocardiography Predicts Long-Term Prognosis in Patients with Acute Myocardial Infarction. Yonsei Med J. 2016 Nov;57(6):1305-6. doi: 10.3349/ymj.2016.57.6.1305. No abstract available. PMID 27593855
- [Background] Bang WD, Kim K, Lee YH, Kwon H, Park Y, Pak HN, Ko YG, Lee M, Joung B. Repolarization Heterogeneity of Magnetocardiography Predicts Long-Term Prognosis in Patients with Acute Myocardial Infarction. Yonsei Med J. 2016 Nov;57(6):1339-46. doi: 10.3349/ymj.2016.57.6.1339. PMID 27593860
- [Background] Motwani M, Dey D, Berman DS, Germano G, Achenbach S, Al-Mallah MH, Andreini D, Budoff MJ, Cademartiri F, Callister TQ, Chang HJ, Chinnaiyan K, Chow BJ, Cury RC, Delago A, Gomez M, Gransar H, Hadamitzky M, Hausleiter J, Hindoyan N, Feuchtner G, Kaufmann PA, Kim YJ, Leipsic J, Lin FY, Maffei E, Marques H, Pontone G, Raff G, Rubinshtein R, Shaw LJ, Stehli J, Villines TC, Dunning A, Min JK, Slomka PJ. Machine learning for prediction of all-cause mortality in patients with suspected coronary artery disease: a 5-year multicentre prospective registry analysis. Eur Heart J. 2017 Feb 14;38(7):500-507. doi: 10.1093/eurheartj/ehw188. PMID 27252451